CLINICAL TRIAL: NCT03303625
Title: A Randomized, Double-blind, Phase 1/2a Study to Evaluate the Safety, Tolerability and Immunogenicity of Ad26.RSV.preF in Adults 18 to 50 Years of Age, RSV-seropositive Toddlers 12 to 24 Months of Age
Brief Title: A Study to Evaluate the Safety, Tolerability and Immunogenicity of an Investigational RSV Vaccine Candidate (Ad26.RSV.preF) in Adults 18 to 50 Years of Age, and RSV-seropositive Toddlers 12 to 24 Months of Age
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CR108371; 2017-001345-27 (EudraCT Number); VAC18194RSV2001 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2017-10-03; First posted 2017-10-06 (Actual); Results first posted 2023-06-23 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Syncytial Viruses; Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort 0: Adults (Ad26.RSV.preF) (Experimental): Participants aged greater than or equal to (>=) 18 to lesser than or equal to (<=) 50 years will receive vector Ad26.RSV.preF at 1*10^11 viral particles (vp) via intramuscular (IM) route (Group 1) on Day 1 and 29.
  Interventions: Biological: Ad26.RSV.preF (1*10^11 vp)
- Cohort 0: Adults (Placebo) (Placebo Comparator): Participants aged >= 18 to <= 50 years will receive placebo via IM route (Group 2) on Day 1 and 29.
  Interventions: Drug: Placebo
- Cohort 1: RSV seropositive Toddlers (Ad26.RSV.preF) (Experimental): RSV seropositive participants aged >=12 to <=24 months will receive Ad26.RSV.preF at 5*10^10 vp via IM route (Group 3) on Day 1 and 29.
  Interventions: Biological: Ad26.RSV.preF (5*10^10 vp)
- Cohort 1: RSV seropositive Toddlers (Placebo) (Placebo Comparator): RSV seropositive participants aged >= 12 to <= 24 months will receive placebo via IM route (Group 4) on Day 1 and 29.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Ad26.RSV.preF (1*10^11 vp) — Participants will receive two doses of 0.5 milliliter (mL) (1*10^11 vp) via IM route on Day 1 and 29 of Ad26.RSV.preF.
  Other Names: JNJ-64400141
  Arms: Cohort 0: Adults (Ad26.RSV.preF)
Biological: Ad26.RSV.preF (5*10^10 vp) — RSV seropositive participants will receive two doses of 0.25 mL (5*10^10 vp) via IM route on Day 1 and 29 of Ad26.RSV.preF.
  Other Names: JNJ-64400141
  Arms: Cohort 1: RSV seropositive Toddlers (Ad26.RSV.preF)
Drug: Placebo — Participants will receive either 0.5 mL (cohort 0) or 0.25 mL (cohort 1) of placebo via IM route on Day 1 and 29.
  Arms: Cohort 0: Adults (Placebo); Cohort 1: RSV seropositive Toddlers (Placebo)

SUMMARY:
The purpose of this study is to assess the safety and tolerability of an intramuscular regimen of two doses (1*10^11 viral particles [vp]) of an investigational respiratory syncytial virus (RSV) vaccine candidate (adenovirus serotype 26 respiratory syncytial virus pre-fusion conformation stabilized F protein [pre-F] [Ad26.RSV.preF]) in adults aged 18 to 50 years and RSV-seropositive toddlers aged 12 to 24 months.

DETAILED DESCRIPTION:
The study, designed to assess the safety and tolerability of two doses given one month apart of Ad26.RSV.preF, an investigational RSV vaccine candidate based on a Ad26 vector expressing the RSV F protein, will be conducted in a double blinded manner. The study will be divided in two sequential cohorts: cohort 0 (18-50 year-old adults) and cohort 1 (12-24 month-old RSV seropositive toddlers). The vaccine safety will be monitored by reporting solicited and unsolicited adverse events (AEs) and all serious adverse events (SAEs). The data will be reviewed by an independent data monitoring committee (IDMC) to assess safety data and to ensure the continuing safety of the participants enrolled in this study. The safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Adults Participants:

* Participant must be in good health, without significant medical illness, on the basis of physical examination, medical history, and vital signs measurement
* Participant must be healthy on the basis of clinical laboratory tests performed at screening. If the results of the laboratory screening tests are outside the local laboratory normal reference ranges and additionally within the limits of toxicity Grade 1 according to the United stated (US) Food and Drug Administration (FDA) toxicity tables, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant and appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* All women of childbearing potential must have a negative highly sensitive serum beta-human chorionic gonadotropin (Beta-hCG) pregnancy test at screening and a negative urine Beta-hCG pregnancy test immediately prior to each study vaccine administration

Pediatric Participants:

* Participant is the product of a normal term pregnancy greater than and equal to (>=) 37 weeks, with a minimum birth weight of 2.5 kilogram (kg)
* Participants must be in good health without any significant medical illness on the basis of physical examination, medical history, and vital signs performed at screening

Exclusion Criteria:

Adults Participants:

* Participant has acute illness (this does not include minor illnesses such as diarrhea) or temperature >=38.0 ºC (degree celsius)/100.4 °F (fahrenheit) within 24 hours prior to the first dose of study vaccine
* Participant has a history of an underlying clinically significant acute or chronic medical condition or physical examination findings for which, in the opinion of the investigator, participation would not be in the best interest of the participant (example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Participant has history of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)

Pediatric Participants:

* Participant's weight is below 10th percentile according to World Health Organization (WHO) pediatric growth and weight charts
* Participant has any clinically significant acute or chronic medical condition that, in the opinion of the investigator, would preclude participation: example, history of seizure disorders, bleeding/clotting disorder, autoimmune disease, active malignancy, systemic infections, congenital heart disease, history of any pulmonary condition requiring medication, atopy, reactive airway disease, medically-confirmed wheezing, bronchoconstriction or treatment with a beta2 agonist, cystic fibrosis, bronchopulmonary dysplasia, chronic pulmonary disease, medically-confirmed apnea, hospitalization for respiratory illness, or mechanical ventilation for respiratory illness

Ages: 12 Months to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2020-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (7):
- Heartland Research Associates, LLC, Newton, Kansas, United States
- Finland (3):
  - Järvenpään rokotetutkimusklinikka, Jarvenpaa
  - University of Tampere/Vaccine Research Center, Tampere
  - University of Tampere/Vaccine Research Center, Turku
- United Kingdom (3):
  - Royal Manchester Children's Hospital, Manchester
  - Oxford Vaccine Group, Oxford
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 0 (Adults): Ad26.RSV.preF: Adult participants aged greater than or equal to (>=) 18 years to less than or equal to (<=) 50 years received a single intramuscular (IM) injection of adenovirus serotype 26 respiratory syncytial virus e pre-fusion conformation stabilized F-protein (Ad26.RSV.preF) at dose of 1*10^11 viral particles (vp) on Day 1 and Day 29.
- Cohort 0 (Adults): Placebo: Adult participants aged >=18 years to <=50 years received a single IM injection of placebo matching to Ad26.RSV.preF (1*10^11 vp) on Day 1 and Day 29.
- Cohort 1 (Toddlers): Ad26.RSV.preF: Respiratory syncytial virus (RSV) seropositive toddler participants aged >=12 to <=24 months received a single IM injection of Ad26.RSV.preF at dose of 5*10^10 vp on Day 1 and Day 29.
- Cohort 1 (Toddlers): Placebo: RSV seropositive toddler participants received a single IM injection of placebo matching to Ad26.RSV.preF (5*10^10 vp) on Day 1 and Day 29.
Period: Overall Study
Arm/Group | Cohort 0 (Adults): Ad26.RSV.preF | Cohort 0 (Adults): Placebo | Cohort 1 (Toddlers): Ad26.RSV.preF | Cohort 1 (Toddlers): Placebo
Started | 8 | 4 | 24 | 12
Completed | 6 | 4 | 24 | 12
Not Completed | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 0 (Adults): Ad26.RSV.preF | Cohort 0 (Adults): Placebo | Cohort 1 (Toddlers): Ad26.RSV.preF | Cohort 1 (Toddlers): Placebo | Total
Number analyzed (Participants) | 8 | 4 | 24 | 12 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 24 | 12 | 36
  Between 18 and 65 years | 8 | 4 | 0 | 0 | 12
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 13 | 8 | 29
  Male | 2 | 2 | 11 | 4 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 4 | 24 | 11 | 45
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  FINLAND | 0 | 0 | 10 | 5 | 15
  UNITED KINGDOM | 8 | 4 | 13 | 6 | 31
  UNITED STATES | 0 | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local Adverse Events (AEs) for 7 Days After First Vaccination
Description: An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with study vaccine. Solicited local AEs were precisely defined events that participants were specifically asked about and which were noted by participants in the diary. Solicited local AEs included erythema, swelling/induration, and pain/tenderness.
Time Frame: For 7 days after first vaccination on Day 1 (Up to Day 7)
Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 0 (Adults): Ad26.RSV.preF | Cohort 0 (Adults): Placebo | Cohort 1 (Toddlers): Ad26.RSV.preF | Cohort 1 (Toddlers): Placebo
Number analyzed (Participants) | 8 | 4 | 24 | 12
Participants | 8 | 1 | 14 | 4

2. Primary Outcome: Number of Participants With Solicited Local Adverse Events (AEs) for 7 Days After Second Vaccination
Description: as for outcome 1
Time Frame: For 7 days after second vaccination on Day 29 (Up to Day 35)
Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study vaccine. Here, 'N' (number of participant analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 0 (Adults): Ad26.RSV.preF | Cohort 0 (Adults): Placebo | Cohort 1 (Toddlers): Ad26.RSV.preF | Cohort 1 (Toddlers): Placebo
Number analyzed (Participants) | 6 | 4 | 24 | 12
Participants | 6 | 0 | 14 | 4

3. Primary Outcome: Number of Participants With Solicited Systemic Adverse Events for 7 Days After First Vaccination
Description: An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with study vaccine. Solicited systemic AEs included were for adult participants: fatigue, headache, myalgia, arthralgia, chills, nausea and fever (defined as body temperature >=38 degree celsius [°C]; for pediatric participants: loss of appetite, vomiting, diarrhea, decreased activity/lethargy, irritability/crying and fever (i.e., body temperature >=38 °C).
Time Frame: For 7 days after first vaccination on Day 1 (Up to Day 7)
Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 0 (Adults): Ad26.RSV.preF | Cohort 0 (Adults): Placebo | Cohort 1 (Toddlers): Ad26.RSV.preF | Cohort 1 (Toddlers): Placebo
Number analyzed (Participants) | 8 | 4 | 24 | 12
Participants | 8 | 1 | 23 | 10

4. Primary Outcome: Number of Participants With Solicited Systemic Adverse Events for 7 Days After Second Vaccination
Description: as for outcome 3
Time Frame: For 7 days after second vaccination on Day 29 (Up to Day 35)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 0 (Adults): Ad26.RSV.preF | Cohort 0 (Adults): Placebo | Cohort 1 (Toddlers): Ad26.RSV.preF | Cohort 1 (Toddlers): Placebo
Number analyzed (Participants) | 6 | 4 | 24 | 12
Participants | 4 | 1 | 22 | 9

5. Primary Outcome: Number of Participants With Unsolicited Adverse Events for 28 Days After First Vaccination
Description: An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with study vaccine. Unsolicited adverse events included all adverse events for which the participant is not specifically questioned in the participant diary.
Time Frame: For 28 days after first vaccination on Day 1 (Up to Day 28)
Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 0 (Adults): Ad26.RSV.preF | Cohort 0 (Adults): Placebo | Cohort 1 (Toddlers): Ad26.RSV.preF | Cohort 1 (Toddlers): Placebo
Number analyzed (Participants) | 8 | 4 | 24 | 12
Participants | 5 | 0 | 11 | 8

6. Primary Outcome: Number of Participants With Unsolicited Adverse Events for 28 Days After Second Vaccination
Description: as for outcome 5
Time Frame: For 28 days after second vaccination on Day 29 (Up to Day 56)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 0 (Adults): Ad26.RSV.preF | Cohort 0 (Adults): Placebo | Cohort 1 (Toddlers): Ad26.RSV.preF | Cohort 1 (Toddlers): Placebo
Number analyzed (Participants) | 6 | 4 | 24 | 12
Participants | 4 | 1 | 12 | 6

7. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with study vaccine. SAE is any untoward medical occurrence that at any dose may result in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product.
Time Frame: From Day 1 (post-vaccination) to end of the study (up to 2 years 4 months)
Population: The safety analysis set included all participants who were randomized and received at least 1 dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 0 (Adults): Ad26.RSV.preF | Cohort 0 (Adults): Placebo | Cohort 1 (Toddlers): Ad26.RSV.preF | Cohort 1 (Toddlers): Placebo
Number analyzed (Participants) | 8 | 4 | 24 | 12
Participants | 0 | 0 | 1 | 2

8. Secondary Outcome: Respiratory Syncytial Virus (RSV) A2 Strain Neutralization Antibody Titers at Days 1, 29, 57 and 211
Description: RSV A2 strain neutralizing antibody titers of the vaccine-induced immune response was assessed through virus neutralization assay.
Time Frame: Day 1 (predose), Post-dose on Days 29, 57 and 211
Population: The Per-protocol Immunogenicity (PPI) set included all randomized and vaccinated participants for whom immunogenicity data were available, excluding participant samples with major protocol deviations expecting to impact the immunogenicity outcomes. Here, 'n' (number analyzed) signifies the number of participants evaluable at a specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Cohort 0 (Adults): Ad26.RSV.preF | Cohort 0 (Adults): Placebo | Cohort 1 (Toddlers): Ad26.RSV.preF | Cohort 1 (Toddlers): Placebo
Number analyzed (Participants) | 8 | 3 | 17 | 9
Titers
  Day 1 (pre-dose) | 329 [252 to 431] | 547 [86 to 3489] | 121 [76 to 191] | 187 [100 to 349]
  Post dose 1: Day 29: number analyzed (Participants) | 6 | 3 | 17 | 7
  Post dose 1: Day 29 | 1089 [483 to 2456] | 603 [101 to 3596] | 1608 [730 to 3544] | 156 [68 to 358]
  Post dose 2: Day 57: number analyzed (Participants) | 6 | 3 | 17 | 8
  Post dose 2: Day 57 | 926 [485 to 1769] | 566 [114 to 2805] | 2235 [1586 to 3150] | 198 [89 to 441]
  Post dose 2: Day 211: number analyzed (Participants) | 6 | 3 | 16 | 7
  Post dose 2: Day 211 | 704 [325 to 1526] | 574 [139 to 2374] | 1164 [734 to 1847] | 165 [70 to 387]

9. Secondary Outcome: Pre-Fusion RSV Fusion Protein (F-protein) Geometric Mean Titers (GMTs) as Assessed by Enzyme-linked Immunosorbent Assay (ELISA) at Days 1, 29, 57 and 211
Description: GMT (ELISA units per liter [EU/L]) of RSV F protein in pre-fusion form as assessed by ELISA was reported.
Time Frame: Pre-fusion on Days 1, 29, 57 and 211
Population: The PPI set included all randomized and vaccinated participants for whom immunogenicity data were available, excluding participant samples with major protocol deviations expecting to impact the immunogenicity outcomes. Here, 'n' (number analyzed) signifies the number of participants evaluable at a specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/L
Arm/Group | Cohort 0 (Adults): Ad26.RSV.preF | Cohort 0 (Adults): Placebo | Cohort 1 (Toddlers): Ad26.RSV.preF | Cohort 1 (Toddlers): Placebo
Number analyzed (Participants) | 8 | 3 | 17 | 9
EU/L
  Day 1 | 197 [132 to 295] | 249 [50 to 1234] | 59 [36 to 97] | 113 [57 to 223]
  Day 29: number analyzed (Participants) | 6 | 3 | 17 | 8
  Day 29 | 441 [304 to 639] | 261 [60 to 1138] | 1174 [524 to 2630] | 106 [56 to 199]
  Day 57: number analyzed (Participants) | 6 | 3 | 17 | 8
  Day 57 | 481 [317 to 729] | 244 [60 to 992] | 1918 [1497 to 2456] | 148 [54 to 402]
  Day 211: number analyzed (Participants) | 6 | 3 | 16 | 7
  Day 211 | 418 [264 to 664] | 292 [45 to 1895] | 924 [639 to 1334] | 120 [39 to 370]

10. Secondary Outcome: Post-Fusion RSV Fusion Protein (F-protein) Geometric Mean Titers (GMTs) as Assessed by ELISA at Days 1, 29, 57 and 211
Description: GMT (ELISA units per liter [EU/L]) of RSV F protein in post-fusion form as assessed by ELISA was reported.
Time Frame: Post-fusion on Days 1, 29, 57 and 211
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: EU/L
Arm/Group | Cohort 0 (Adults): Ad26.RSV.preF | Cohort 0 (Adults): Placebo | Cohort 1 (Toddlers): Ad26.RSV.preF | Cohort 1 (Toddlers): Placebo
Number analyzed (Participants) | 8 | 3 | 17 | 9
EU/L
  Day 1 | 196 [112 to 346] | 191 [19 to 1879] | 77 [48 to 125] | 94 [46 to 190]
  Day 29: number analyzed (Participants) | 6 | 3 | 17 | 8
  Day 29 | 328 [207 to 521] | 207 [25 to 1738] | 686 [371 to 1268] | 86 [47 to 158]
  Day 57: number analyzed (Participants) | 6 | 3 | 17 | 8
  Day 57 | 341 [198 to 589] | 179 [23 to 1370] | 863 [630 to 1184] | 109 [52 to 232]
  Day 211: number analyzed (Participants) | 6 | 3 | 16 | 7
  Day 211 | 268 [142 to 507] | 181 [18 to 1870] | 420 [306 to 576] | 91 [33 to 256]

11. Secondary Outcome: Percentage of Cytokine Subsets (CD4, CD8, Th1 and Th2 Cytokines) to Evaluate Total Cytokine Response at Days 1, 29 and 57
Description: Total cytokine response (CD4, CD8, Th1 and Th2 Cytokines) after in vitro RSV F protein peptide stimulation was reported as the percentage of CD4+ and CD8+ T cells that produce at least 1 of 3 cytokines.
Time Frame: Day 1 (predose) and Post-dose on Days, 29, and 57
Population: PPI set: all randomized and vaccinated participants for whom immunogenicity data were available, excluding participant samples with major protocol deviations expecting to impact immunogenicity outcomes. 'N' (number of participants analyzed)=number of participants who were evaluable for this outcome measure, 'n' (number analyzed)=number of participants evaluable at specified timepoint and '0' in number analyzed field=none of participants were applicable for evaluation at specified time point.
Measure: Median (Inter-Quartile Range); unit: Percentage of cytokine cell subsets
Arm/Group | Cohort 0 (Adults): Ad26.RSV.preF | Cohort 0 (Adults): Placebo | Cohort 1 (Toddlers): Ad26.RSV.preF | Cohort 1 (Toddlers): Placebo
Number analyzed (Participants) | 4 | 3 | 14 | 8
Percentage of cytokine cell subsets
  CD4: Day 1: number analyzed (Participants) | 4 | 3 | 13 | 8
  CD4: Day 1 | 0.058 [0.057 to 0.067] | 0.054 [0.048 to 0.108] | 0.030 [0.013 to 0.095] | 0.050 [0.015 to 0.079]
  CD4: Day 29: number analyzed (Participants) | 3 | 3 | 13 | 8
  CD4: Day 29 | 0.168 [0.100 to 0.210] | 0.058 [0.051 to 0.082] | 0.089 [0.062 to 0.131] | 0.074 [0.056 to 0.123]
  CD4: Day 57: number analyzed (Participants) | 4 | 3 | 0 | 0
  CD4: Day 57 | 0.148 [0.115 to 0.351] | 0.039 [0.024 to 0.116] |  |
  CD8: Day 1: number analyzed (Participants) | 4 | 3 | 13 | 8
  CD8: Day 1 | 0.041 [0.033 to 0.084] | 0.075 [0.005 to 0.141] | 0.033 [0.024 to 0.049] | 0.041 [0.025 to 0.081]
  CD8: Day 29: number analyzed (Participants) | 3 | 3 | 14 | 8
  CD8: Day 29 | 0.145 [0.080 to 0.233] | 0.092 [0.022 to 0.105] | 0.077 [0.024 to 0.116] | 0.053 [0.016 to 0.110]
  CD8: Day 57: number analyzed (Participants) | 4 | 3 | 0 | 0
  CD8: Day 57 | 0.081 [0.070 to 0.211] | 0.062 [0.003 to 0.185] |  |
  Th1: Day 1: number analyzed (Participants) | 4 | 3 | 13 | 8
  Th1: Day 1 | 0.045 [0.028 to 0.065] | 0.054 [0.031 to 0.096] | 0.007 [0.003 to 0.022] | 0.018 [0.011 to 0.027]
  Th1: Day 29: number analyzed (Participants) | 3 | 3 | 13 | 8
  Th1: Day 29 | 0.098 [0.040 to 0.146] | 0.049 [0.037 to 0.057] | 0.034 [0.025 to 0.078] | 0.028 [0.017 to 0.055]
  Th1: Day 57: number analyzed (Participants) | 4 | 3 | 0 | 0
  Th1: Day 57 | 0.112 [0.083 to 0.302] | 0.039 [0.008 to 0.061] |  |
  Th2: Day 1: number analyzed (Participants) | 4 | 3 | 13 | 8
  Th2: Day 1 | 0.006 [0.001 to 0.016] | 0.001 [0.001 to 0.002] | 0.002 [0.001 to 0.004] | 0.004 [0.001 to 0.005]
  Th2: Day 29: number analyzed (Participants) | 3 | 3 | 13 | 8
  Th2: Day 29 | 0.003 [0.002 to 0.006] | 0.001 [0.001 to 0.001] | 0.005 [0.001 to 0.007] | 0.003 [0.002 to 0.007]
  Th2: Day 57: number analyzed (Participants) | 4 | 3 | 0 | 0
  Th2: Day 57 | 0.003 [0.001 to 0.022] | 0.001 [0.001 to 0.001] |  |

ADVERSE EVENTS:
Time Frame: From Day 1 (post-vaccination) up to end of the study (up to 2 years 4 months)
Description: The safety analysis set included all participants who were randomized and received at least 1 dose of study vaccine.
Arm/Group | Cohort 0 (Adults): Ad26.RSV.preF | Cohort 0 (Adults): Placebo | Cohort 1 (Toddlers): Ad26.RSV.preF | Cohort 1 (Toddlers): Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/4 | 0/24 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/4 | 1/24 | 2/12
Other Adverse Events (participants affected / at risk) | 6/8 | 1/4 | 19/24 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 0 (Adults): Ad26.RSV.preF (N=8) | Cohort 0 (Adults): Placebo (N=4) | Cohort 1 (Toddlers): Ad26.RSV.preF (N=24) | Cohort 1 (Toddlers): Placebo (N=12)
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 0 (Adults): Ad26.RSV.preF (N=8) | Cohort 0 (Adults): Placebo (N=4) | Cohort 1 (Toddlers): Ad26.RSV.preF (N=24) | Cohort 1 (Toddlers): Placebo (N=12)
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Teething (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Influenza Like Illness (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Allergy to Animal (Immune system disorders) | 0 | 0 | 0 | 1
Anal Infection (Infections and infestations) | 0 | 0 | 1 | 0
Body Tinea (Infections and infestations) | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0
Enterovirus Infection (Infections and infestations) | 0 | 0 | 0 | 1
Hand-Foot-And-Mouth Disease (Infections and infestations) | 0 | 0 | 1 | 0
Oral Herpes (Infections and infestations) | 0 | 0 | 1 | 0
Otitis Externa (Infections and infestations) | 1 | 0 | 0 | 0
Otitis Media (Infections and infestations) | 0 | 0 | 4 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 4 | 4
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Skin Bacterial Infection (Infections and infestations) | 0 | 0 | 1 | 0
Tinea Infection (Infections and infestations) | 0 | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 0 | 8 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 1 | 0
Viral Rash (Infections and infestations) | 0 | 0 | 0 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 2
Heart Rate Increased (Investigations) | 1 | 0 | 0 | 0
Influenza B Virus Test Positive (Investigations) | 1 | 0 | 0 | 0
Lymphocyte Count Decreased (Investigations) | 1 | 0 | 0 | 0
Respiratory Syncytial Virus Test Positive (Investigations) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0
Loss of Consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 2
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory Tract Irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/25/NCT03303625/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-25): https://cdn.clinicaltrials.gov/large-docs/25/NCT03303625/SAP_001.pdf